CLINICAL TRIAL: NCT05060094
Title: Comparison of Outcomes Between Single-step Transepithelial Photorefractive Keratectomy and Off-flap Epipolis Laser in Situ Keratomileusis
Brief Title: Comparison of Outcomes Between TransPRK and Off-flap Epi-LASIK
Status: Completed | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, director of cataract department, Wenzhou Medical University
Other Study IDs: outcomes of TransPRK
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Refractive Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To compare the quantitative and qualitative optical outcomes between single-step transepithelial photorefractive keratectomy (TransPRK) and off-flap epipolis laser in situ keratomileusis (Epi-LASIK) in moderate to high myopia.we included patients with moderate to high myopia who were randomized to have TransPRK in one eye and Epi-LASIK in the other eye. All patients underwent comprehensive ophthalmological examinations, including uncorrected (UDVA) and corrected distance visual acuities (CDVA), manifest refraction, intraocular pressure, anterior and posterior segment examination, corneal topography measured by Scheimpflug scanning-slit topographer (Pentacam, Oculus Optikgerate GmbH), contrast sensitivity (CS) under photopic and mesopic conditions (CSV-1000E, Vector Vision Inc., Greenville, OH, USA) with correction by spectacles, ocular wavefront aberrometry (OPD-Scan II, Nidek Co. Ltd). At each follow-up, CS and aberration measures were repeated 3 times and the average value was analyzed. Optical parameters were repeated 1, 3, 6, and 12 months after surgery.Statistical analysis was performed using SPSS software (version 22.0, SPSS, Chicago, Inc.). Kolmogorov-Smirnov test was used to check the normal distribution of variables. Student t-test or Wilcoxon rank sum test was used based on the normality of data. A P value less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* corrected distance visual acuity (CDVA) in logarithm of minimal angle of resolution (LogMAR) of 0.10 or better
* refractive error stabilized for at least 1 year
* discontinued contact lens use for at least 2 weeks

Exclusion Criteria:

* presence of corneal scars
* keratoconus
* glaucoma
* retinal diseases
* a history of corneal or intraocular surgery

Ages: 19 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: people accepted refractive surgery
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
aberrations | 2016.03.01-2018.06.05
  ocular high-order aberrations including spherical, coma and trefoil aberrations were measured by OPD-Scan II

SECONDARY OUTCOMES:
contrast sensitivity | 2016.03.01-2018.06.05
  contrast sensitivity and contrast sensitivity under glare condition measurements were performed by the CSV-1000E which could test four spatial frequencies: 3,6,12 and 18 cycles/degree (cpd) at 2.5m. The contrast sensitivity was measured under photopic (596.7cd/㎡) and scotopic (0.01cd/㎡) conditions and the contrast sensitivity under glare condition was taken under scotopic condition with glare
haze | 2016.03.01-2018.06.05
  Corneal haze grade was recorded according to Fantes's report: 0, no haze; 0.5, trace haze only could be seen by oblique illumination; 1,more visible haze not interfering with the visibility of iris details; 2, mild influence of iris details; 3, moderate influence of iris details; 4, marked haze obscuring the stroma of ablation area.
postoperative pain | 2016.03.01-2018.06.05
  Subjective pain scores were evaluated on the third day according to a predetermined scale ranging from 0 to 5 as follows: 0, no pain or discomfort; 1, photophobia and tears; 2, photophobia and tears with mild pain; 3, photophobia and tears with moderate pain that does not require oral medication; 4, photophobia and tears with severe pain that oral medication can relieve; 5, photophobia and tears with severe pain that oral medication cannot relieve.

REFERENCES:
- [Derived] Zhang Y, Li T, Li Z, Dai M, Wang Q, Xu C. Clinical outcomes of single-step transepithelial photorefractive keratectomy and off-flap epipolis-laser in situ keratomileusis in moderate to high myopia: 12-month follow-up. BMC Ophthalmol. 2022 May 23;22(1):234. doi: 10.1186/s12886-022-02443-6. PMID 35606707